CLINICAL TRIAL: NCT04611763
Title: Effect of Preemptive Analgesia With Flurbiprofen Axetil on Perioperative Sleep Quality and Postoperative Pain in Patients Undergoing Laparoscopic Gynecological Surgery.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Flurbiprofen axetil
Record Dates: First submitted 2020-10-29; First posted 2020-11-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Flurbiprofen Axetil; Preemptive Analgesia; Postoperative Pain; Perioperative Sleep Quality; Postoperative Inflammatory Markers
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre FA Group (Experimental)
  Interventions: Drug: Flurbiprofen axetil preoperatively
- Post FA Group (Active Comparator)
  Interventions: Drug: Flurbiprofen axetil postoperatively

INTERVENTIONS:
Drug: Flurbiprofen axetil preoperatively — give Flurbiprofen axetil 15 min before surgery
  Arms: Pre FA Group
Drug: Flurbiprofen axetil postoperatively — give Flurbiprofen axetil at the end of surgery
  Arms: Post FA Group

SUMMARY:
In humans and animals, circadian rhythm sleep cycle is an important function to maintain and regulate basic physiological homeostasis, such as cognitive function, glucose metabolism, memory consolidation, immune function and growth hormone secretion. The induction of general anesthesia leads to a state of reduced responsiveness, which is often described by anesthesiologists and patients as "sleep". However, previous studies have shown that in the case of patients under general anesthesia, besides surgery trauma and general anesthetics may change sleep function and sleep cycle perioperatively, the postoperative complications such as pain, nausea and vomitting etc after general anesthesia may also reduce postoperative sleep quality.Meanwhile, there is a mixed literature linking sleep and markers of systemic inflammation that greater sleep disturbances were associated with higher levels of circulating IL-6 and CRP but not TNF-α. And the effects of inflammatory cytokines may also cause changes in sleep patterns. Flurbiprofen axetil is a new non-steroidal anti infection analgesic(NSAIDs), which is widely used for analgesia to reduce the dose of opioids. It not only has a high affnity for infammatory tissues to achieve targeted drug therapy and prolonged duration of action, but causes analgesia effect through decreasing the biological production of prostaglandins, reducing the reactivity of peripheral nerves to endogenous infammatory factors, and inhibiting the sensitization of central as well as peripheral nervous systems.Furthermore, it could also inhibite the occurrence of adverse reactions, such as declined sleep quality, respiratory depression, nausea and vomiting. Preemptive analgesia is an analgesic intervention that begins before surgery to prevent the nervous system from becoming sensitive to subsequent stimuli that may aggravate pain. A large number of experimental studies have shown that the use of local anesthetics and/or analgesics in advance can prevent central nervous system hyperplasia, thereby reducing postoperative pain. The aim of our study was to investigate the effect of preemptive analgesic with flurbiprofen axetil on postoperative pain, inflammatory markers and sleep quality among patients under general anesthesia. We hypothesized that use flurbiprofen axetil preoperatively would effectively relieve postoperative pain, inhibite inflammtory reaction and improve postoperative sleep quality.

ELIGIBILITY:
Inclusion Criteria:

age: 18-75 ASA: I-II Receive operation under general anesthesia

Exclusion Criteria:

* ①Patients with mental illness;

  * Severe sleep disorders in the past;

    * A history of taking opioids;

      * Patients who are allergic to the drug

        * Patients who have difficulty communicating and refuse to participate in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Postoperative 24 hours pain score | 24 hours after surgery
  Use VAS to evaluated postoperative pain score
perioperative inflammatory markers | the day before surgery
  The inflammtory markers such as system inflammation Index (SII), neutrophil-to-lymphocyte ratio (NLR), and monocyte-to-lymphocyte ratio (MLR) were recorded before and after surgery. SII= platelet count × neutrophil count/lymphocyte count, NLR= neutrophil count/lymphocyte count, MLR= monocyte count/lymphocyte count.
perioperative inflammatory markers | first day after surgery
  The inflammtory markers such as system inflammation Index (SII), neutrophil-to-lymphocyte ratio (NLR) and monocyte-to-lymphocyte ratio (MLR) were recorded before and after surgery. SII= platelet count × neutrophil count/lymphocyte count, NLR= neutrophil count/lymphocyte count, MLR= monocyte count/lymphocyte count.
perioperative inflammatory markers | third day after surgery
  The inflammtory markers such as system inflammation Index (SII), neutrophil-to-lymphocyte ratio (NLR), and monocyte-to-lymphocyte ratio (MLR) were recorded before and after surgery. SII= platelet count × neutrophil count/lymphocyte count, NLR= neutrophil count/lymphocyte count, MLR= monocyte count/lymphocyte count.

SECONDARY OUTCOMES:
preoperative sleep quality | the first night before surgery
  evaluate postoperative sleep quality at the first night before surgery
postoperative sleep quality | the first night after surgery
  evaluate postoperative sleep quality at the first night after surgery
postoperative sleep quality | the third night after surgery
  evaluate postoperative sleep quality at the third night after surgery
postoperative adverse effects | 24 hours after surgery
  evaluate postoperative adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- beijing friendship hospital of Capital Medical university, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang X, Wei W, Leng Z, Song B, Fu M, He J, Zhu J. Preemptive flurbiprofen axetil for sleep-pain-inflammation modulation after laparoscopic gynecological surgery: a prospective, parallel-group randomized controlled trial. Front Pharmacol. 2025 Oct 7;16:1659179. doi: 10.3389/fphar.2025.1659179. eCollection 2025. PMID 41126955